CLINICAL TRIAL: NCT00394407
Title: Comparative Trial Between Insulin Glargine Plus Supplemental Glulisine (Apidra) Versus Sliding Scale Regular Insulin In Hospitalized Patients With Type 2 Diabetes
Brief Title: Basal/Bolus Versus Sliding Scale Insulin In Hospitalized Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry); University of Miami (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 419-2005; 419-2005 (Other: Other)
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Hyperglycemia
Keywords: inpatient; diabetes management; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sliding scale regular insulin (Active Comparator): sliding scale insulin given acqhs
  Interventions: Drug: sliding scale regular insulin
- glargine insulin and glulisine insulin (Active Comparator): glargine basal insulin once a day with prandial glulisine insulin tid
  Interventions: Drug: glargine basal insulin and glulisine prandial insulin

INTERVENTIONS:
Drug: sliding scale regular insulin — SSRI acqhs
  Other Names: Novolin-R
  Arms: sliding scale regular insulin
Drug: glargine basal insulin and glulisine prandial insulin — glargine insulin once a day and glulisine insulin three times a day as long as patient eating
  Other Names: Lantus inuslin, Apidra insulin
  Arms: glargine insulin and glulisine insulin

SUMMARY:
High blood glucose levels in hospitalized patients with diabetes are associated with increased risk of medical complications. Improved glucose control with insulin injections may improve clinical outcome and prevent some of the hospital complications. It is not known; however, what is the best insulin regimen in hospitalized patients. The use of repeated injections of regular insulin (known as sliding scale regimen) is one of the most commonly used insulin regimen for glucose control in hospitalized patients with diabetes. Recently, the combination of basal and rapid acting insulins has been shown to improve glucose control with lower rate of hypoglycemia (low blood sugar).

DETAILED DESCRIPTION:
This study will compare how well regular insulin will compare to glargine (Lantus®) once daily plus glulisine (Apidra®) insulin before meals in hospitalized patients with type 2 diabetes and elevated blood glucose (sugar) levels. Lantus is a long-acting insulin which is given subcutaneously (under the skin) once daily. Apidra is a rapid-acting insulin which is given subcutaneously several times a day and frequently before meals. Regular insulin is a short-acting insulin in clinical use for more than 20 years that is also given subcutaneously several times per day. Lantus, Apidra and regular insulins are approved for use in the treatment of patients with diabetes by the FDA.

This investigator-initiated research will be conducted at Grady Memorial Hospital, Atlanta and at Jackson Memorial Hospital, Miami. Dr. Umpierrez designed the study and will serve as principal investigator. A total of 65 patients will be recruited at Grady and 65 patients at the Jackson Memorial Hospital. This study is supported by Sanofi-Aventis Pharmaceuticals.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 70 years admitted to a general medicine service.
2. A known history of type 2 diabetes mellitus > 3 months, receiving either diet alone or any combination of oral antidiabetic agents (sulfonylureas, metformin, thiazolidinediones).
3. Subjects must have an admission blood glucose > 140 mg and < 400 mg/dL without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 mEq/L or positive serum or urinary ketones).

Exclusion Criteria:

1. Subjects with increased blood glucose concentration, but without a known history of diabetes.
2. Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria [57].
3. Patients with known HIV, acute critical or surgical illness and/or expected to require admission to a critical care unit (ICU, CCU), corticosteroid therapy, or to undergo surgery during the hospitalization course.
4. Patients with clinically relevant hepatic disease or impaired renal function, as shown by a serum creatinine ≥3.0.
5. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
6. Patients with recognized or suspected endocrine disorders associated with increased insulin resistance, acromegaly, or hyperthyroidism.
7. Female subjects are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
blood glucose control | During hospitalization
  Differences in BG control will be assessed between the 2 arms acqhs and as needed for those patients hospitalized on the non-medical floors

SECONDARY OUTCOMES:
frequency of hypoglycemia | during the hospitalization
  assess differences in the frequency of hypoglycemia between the 2 study arms
frequency of severe hyperglycemia (BG > 400 mg/dl), | during the hospitalization
  evaluate differences in severe hyperglycemia between the 2 study arms
length of hospital stay | during hospitalization
  differences in LOS between study arms
inflammatory markers | during hospitalization
  C-reactive protein, interleukin-6, and tumor necrosis factor

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- University of Miami School of Medicine, Coral Gables, Florida, United States

REFERENCES:
- [Derived] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708